CLINICAL TRIAL: NCT04901416
Title: An Open-Label Pilot Study to Evaluate the Safety and Efficacy of DVX201 NK Cells in Patients With Relapsed or Refractory AML or High Risk MDS or High Risk Overlapping Myelodysplastic / Myeloproliferative Neoplasms
Brief Title: Safety and Efficacy of Allogeneic NK Cell Infusions in Patients With Relapsed/Refractory AML and High Risk MDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Coeptis Therapeutics (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DVX201-AML-01
Record Dates: First submitted 2021-05-21; First posted 2021-05-25 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-04

CONDITIONS: AML, Adult Recurrent; MDS
Keywords: NK cells; AML; Allogeneic; MDS; Relapse
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Intervention Model Description: This is a single arm, unblinded, non-randomized Phase 1 dose-finding study of DVX201.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): 1. Lymphodepleting (LD) chemotherapy will be administered daily for 3 days to all subjects prior to DVX201. Lymphodepleting chemotherapy will consist of the following:
     1. Cyclophosphamide 300 mg/m2 IV over 30 to 60 minutes daily x 3 (day -5 to day - 3)
     2. Fludarabine 30 mg/m2 IV over 30 minutes daily x 3 (day -5 to day -3)
  2. Patients will receive DVX201 at one of 3 prespecified doses infused on day 0 and 7 (± 1 day) for 1 cycle.
  Interventions: Biological: DVX201

INTERVENTIONS:
Biological: DVX201 — Based upon the occurrence of DLT (does limiting toxicity), the MTD will be estimated as the highest dose at which the toxicity probability is the closest to the target probability (denoted pT=0.30) following up to 2 doses of DVX201. The corresponding dose allocation methodology is a modified toxicity interval design based upon (Ji et al., 2010; Ji et al., 2013).
  All patients who have at least one dose initiated will be included in the safety analysis. Patients who are enrolled but never exposed to investigational product will be replaced for all analyses. Patients who get exposed to lymphodepleting chemotherapy will be followed and reported for outcomes overall, but for determination of safety and efficacy, only those subjects who have been exposed to the investigational agent will be included.

SUMMARY:
This study involves the use of an investigational cell therapy known as DVX201. DVX201 is an investigational cell therapy that contains a type of white blood cell called natural killer (NK) cells. NK cells are a normal part of your immune system and have a lifespan of only about two weeks. They are called natural killer cells because they have the natural ability to identify and kill cells in the body that are abnormal, like cancer cells or virally infected cells. But fighting cancer can also lead to exhaustion and abnormal function of NK cells. It can also result in a significant decrease in the number of NK cells in the blood, making it more difficult for the immune system to control the disease. We believe that infusion of healthy, functional NK cells into patients with AML or MDS may boost the immune system and help by killing cancer cells that remain after chemotherapy. DVX201 is an investigational NK cell therapy that may provide a rapid and temporary source of healthy NK cells that are better able to fight those cancer cells.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age and weighing at least 40 kg, inclusive, with persistence or relapse/progression of AML, MDS, or MDS/MPN overlap (within 28 days of enrollment) and:

   1. a diagnosis of persistence or relapse/progression of AML and ≥ 5% blasts in the marrow or blood following at least 1 cycle of induction therapy, or
   2. a diagnosis of intermediate, high, or very high-risk MDS according to IPSS-R classification (Greenberg et al., 2012) who are resistant or refractory to at least one course of therapy including demethylating agents (having had at least 4 cycles) with ≥ 5% blasts in the marrow or blood, or
   3. a diagnosis of overlap of an MPN with MDS features and also are resistant or refractory to at least one course of therapy including demethylating agents (having had at least 4 cycles) with ≥ 5% blasts in the marrow or blood.
2. Written informed consent in accordance with federal, local, and institutional guidelines.
3. Must be able to adhere to the study visit schedule and other protocol requirements.
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Meet the following laboratory criteria within 7 days of enrollment:

   1. ALT/SGPT and AST/SGOT < 3x the upper limit of normal (ULN) unless due to underlying disease state
   2. Calculated creatinine clearance ≥ 45.0 mL/min as estimated by Cockcroft Gault and dialysis independent (Cockcroft et al., 1976)
   3. Total bilirubin ≤ 2.0 mg/dL (Patients with Gilbert's or Meulengracht Syndrome must have a total bilirubin < 5.0 mg/dL).
6. Females cannot be pregnant or breast-feeding from time of enrollment or for 3 months post final infusion.
7. Women of childbearing potential is willing to use 2 highly effective methods of contraception while receiving study treatment and for an additional 3 months after the last dose of protocol-specified therapy. Men who have a female partner of childbearing potential are together willing to use 2 highly effective forms of contraception for at least an additional 3 months after the last dose of protocol- specified therapy.
8. Patients status post allogeneic BMT or other donor lymphocyte infusions are eligible, but they must be at least 60 days from the last infusion of cell therapy products.
9. Patients must have other anti-leukemia therapies stopped 2 weeks prior to infusion on this study. Hydroxyurea and/or pheresis ARE allowed prior to this study until 1 day prior to infusion.

Exclusion Criteria:

1. Weight less than 40 kg.
2. Patients with progressive infections at time of first infusion (patients with treated infections documented as controlled by the treating team are eligible).
3. Patients with history of active seizure disorder (having a documented seizure within the prior year) or any autoimmune disease with CNS involvement.
4. Major surgery, chemotherapy, systemic therapy (excluding hydroxyurea, steroids, and any targeted small molecules or biologics), or radiotherapy within 14 days or 5 half-lives (whichever is shorter) prior to Cycle 1.
5. Patients with proven, progressive severe autoimmune disease such as multiple sclerosis, active Guillain Barré syndrome, poliomyelitis, Sjogren's are not eligible.

   Given the immediate, life threatening nature of the relapsed cancer in this patient population, those with other stable and non-immediate non-threatening autoimmune disorders (such as thyroid disease or diabetes and others) are eligible.
6. Diagnosis of any other malignancy within 3 years, except for adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the breast or of the cervix, low grade prostate cancer on surveillance without any plans for treatment intervention other than hormonal therapy, or prostate cancer that has been adequately treated with prostatectomy or radiotherapy and currently with no evidence of disease or symptoms.
7. Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism.
8. Any active acute Graft-versus-Host Disease (GvHD) > Grade 1 overall or systemic treatment of more than 10 mg prednisone daily (or equivalent); patients must have been off any calcineurin inhibitors for at least 28 days prior to starting therapy on this study.
9. Current use of immunosuppressive medications at the time of study enrollment and within 2 weeks of any study treatments, except:

   1. Intranasal, inhaled, topical steroids, or local steroid injection
   2. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent
   3. Steroids as premedication for hypersensitivity reactions at physiologic doses ≤ 10 mg/day of prednisone or equivalent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities | Through 28 days post second infusion of ccell therapy (DVX201)
  Dose limiting toxicities include toxicities with cell therapy infusion, CRS, organ toxicity, GVHD as defined in the protocol

SECONDARY OUTCOMES:
Disease response | through approximately 30 days post second cell therapy infusion (DVX201)
  Patient's response to DVX201 as CR, CRi, PR, MLFS, PD, or NR based on the Investigator's evaluation using standardized NCCN criteria
Duration of response | Through study completion, an average of 6 months start of therapy
  Patients with disease response will be followed to see how long the duration of this response is and if primary disease recurs or worsens

OTHER OUTCOMES:
Length of time that DVX201 (NK cells) remain in the blood | through 28 days post second infusion of DVX201
  Evaluation of persistence of DVX201 in the peripheral blood by chimerism testing
1. Evaluation of NK cells in blood samples after DVX201 infusion to look for markers of NK cell exhaustion and activation | through 28 days post second infusion of DVX201
  Characterization of circulating NK and other immune cells in the peripheral blood by flow immunophenotyping

CONTACTS AND LOCATIONS:
Overall Officials: David A Rizzieri, MD, Study Chair — Novant Health; Thomas W LeBlanc, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States